CLINICAL TRIAL: NCT02366221
Title: Upper-Extremity Bone or Joint Surgery: Long Term Outcome
Status: Enrolling by invitation | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Neal Chung-Jen Chen, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 1999P008705
Record Dates: First submitted 2014-10-16; First posted 2015-02-19 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Upper Extremity Fractures; Upper Extremity Non-Fracture Bone and Joint Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All subjects: Subjects with a history of complex arm trauma
  Interventions: Other: 60-minute visit to the outpatient clinic; Other: Phone Interview

INTERVENTIONS:
Other: 60-minute visit to the outpatient clinic — An interview, an injury-specific physical exam and/or a set of xrays.
Other: Phone Interview — If subject cannot return to office in Boston, researcher may conduct interview over the phone.

SUMMARY:
The specific aim of the study is to obtain long-term follow-up information on patients who have completed their standard clinical care in the Orthopaedic Hand and Upper Extremity Service. The study will help to qualify and quantify long-term recovery and outcomes from uncommon upper extremity fractures, as well as non-fracture bone and joint conditions. The hypotheses vary, but generally focus on the patterns of injury, the results of treatment and the complications encountered.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of complex arm or leg trauma who have completed their normal care in the Orthopaedic Hand and Upper Extremity Service

Exclusion Criteria:

* Vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a history of complex arm or leg trauma who have completed their normal care in the Orthopaedic Hand and Upper Extremity Service
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 1998-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | 5 years (expected average)
  Range of motion of joints measured in degrees with goniometer

SECONDARY OUTCOMES:
Upper Extremity Function | 5 years (expected average)
  PROMIS (Patient Reported Outcomes Measurement Information Systems) Upper Extremity Questionnaire
Pain Interference | 5 years (expected average)
  PROMIS Pain Interference Questionnaire
Depression | 5 years (expected average)
  PROMIS Depression Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Neal Chen, MD, Principal Investigator — Massachusetts General Hospital